CLINICAL TRIAL: NCT05278832
Title: A Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of QLS31905 in Patients With Claudin18.2-positive Advanced Solid Tumors
Brief Title: A Study of QLS31905 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS31905-101
Record Dates: First submitted 2022-02-23; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS31905 (Experimental): QLS31905 injection
  Interventions: Drug: QLS31905

INTERVENTIONS:
Drug: QLS31905 — QLS31905 injection

SUMMARY:
This is a multi-center, open-label design to evaluate the safety and tolerance of QLS31905 in patients with advanced solid tumors, together with an assessment of pharmacokinetic characteristics and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. ≥18 years.
3. Female or male.
4. ECOG performance status score 0 or 1.
5. Histologically or cytologically confirmed diagnosis of advanced solid tumors.
6. Adequate haematological, hepatic and renal function.

Exclusion Criteria:

1. Any anticancer therapy or immunotherapy within 4 weeks prior to the start of study treatment.
2. Untreated or symptomatic central nervous system (CNS) metastases or leptomeningeal disease.
3. Patients with a history of monoclonal antibody allergic reaction.
4. Known human immunodeficiency virus infection or known symptomatic hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities(DLTs) | 2 years
  Number of participants experiencing DLTs According to NCI-CTCAE v.5.0，To evaluate the safety and tolerability of QLS31905
Maximum tolerated Dose(MTD) | 2 years
  To evaluate the safety and tolerability of QLS31905

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 2 years
  Progression free survival will be determined from investigator derived tumor assessments per RECIST 1.1.
Objective response rate (ORR) | 2 years
  Objective Response Rate (ORR) is the percentage of CR+PR
Disease control rate (DCR) | 2 years
  Disease control Rate (DCR) is the percentage of CR+PR+SD
adverse events (AE) | 2 years
  To evaluate the safety and tolerability of QLS31905
Cmax | 2 years
  Maximum concentration (Cmax) of the drug after administration
AUC | 2 years
  The area under the curve (AUC) of serum concentration of the drug after the administration

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China